CLINICAL TRIAL: NCT03586518
Title: Validating the Accuracy of Novel, Non-contrast, Cardiac Magnetic resOnaNce Imaging in Defining Myocardial FIbRosis in Patients With End-stage Renal Disease on haeModialysis: the CONFIRM Study
Brief Title: Validating Novel, Non-contrast Cardiac MRI Imaging in Haemodialysis Patients
Acronym: CONFIRM
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 0674
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: End Stage Kidney Disease; Fibrosis Myocardial
Keywords: Cardiac MRI; Hemodialysis; Myocardial Fibrosis; Myocardial Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Myocarditis | interventions — Echocardiography; Electrocardiography, Ambulatory; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient hearts explanted post-mortem
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haemodialysis patients: The plans for patient recruitment were developed in partnership with our local haemodialysis patient participation and involvement group. Patients will be identified from the supportive care register established for haemodialysis patients in Leicester in 2008.
  Inclusion:
  * Prevalent haemodialysis patient (more than 3 months)
  * Active on the supportive care register with anticipated death in the subsequent 12 months
  * Able to give informed consent
  * Consent to donation of heart for research following death
  * Able to understand written and verbal explanations in English
  Exclusion:
  * Contraindication to MRI scan (e.g. pacemaker, incompatible metallic implants, claustrophobia)
  * Patients with expected or potential infiltrative cardiomyopathy (e.g. amyloidosis)
  * Unable to give informed consent
  * Unable to understand written and verbal explanations in English
  Interventions: Diagnostic Test: Cardiac MRI scan; Diagnostic Test: Echocardiogram; Procedure: Cardiac explantation; Diagnostic Test: 48-Hour continuous cardiac monitoring; Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Cardiac MRI scan — A non-contrast cardiac MRI (CMR) scan at 3-Tesla platform (Skyra, Siemens Medical Imaging, Erlangen, Germany).
  This non-contrast CMR scan will principally determine: Left ventricular (LV) mass and volumes/ejection fraction and; fibrosis using T1 mapping.
  Other Names: CMR
Diagnostic Test: Echocardiogram — Assessments will include: LV size and function as per the American Society of Echocardiography guidelines. In addition specific focus will be paid end-diastolic integrated backscatter measurements.
  Other Names: ECHO
Procedure: Cardiac explantation — A limited post-mortem will be performed to retrieve patients' hearts for preparation and storage at St George's University, London where direct comparison will be made between levels of scarring seen directly under the microscope between that on the MRI scans.
Diagnostic Test: 48-Hour continuous cardiac monitoring — Attach continuous Holter monitor (Schiller, medilog®AR12 plus/AR4 plus/FD5 plus, Baar, Switzerland) that will start before dialysis and terminate just before the subsequent dialysis treatment 48h later.
  Other Names: Holter
Diagnostic Test: Blood samples — Collect blood samples from the arterial needle before dialysis. Approximately 30 millilitres of blood will be collected and then be pipetted into cryotubes and frozen at -80°C in an electronically monitored freezer for analysis in batches throughout the study. These samples will be used to investigate the relationship between circulating biomarkers of fibrosis, the MRI scans and the histological samples.

SUMMARY:
There are currently no good ways of measuring levels of scarring in the hearts of patients with advanced kidney disease and patients on dialysis, although recent research has shown a new cardiac MRI technique, called native T1 mapping, may provide a solution to this. To assess the accuracy of this novel technique in dialysis patients, it is essential to undertake a study which compares native T1 mapping to actual levels of scarring in the hearts of patients on dialysis.

DETAILED DESCRIPTION:
Native T1 mapping is a novel, non-contrast, cardiac MRI technique that characterises myocardial tissue by exploiting the different water content of tissues. It correlates well with histo-pathological levels of myocardial fibrosis in diseases of pressure overload such as aortic stenosis. There is growing evidence to demonstrate the potential of native T1 mapping as an imaging biomarker of myocardial fibrosis in patients with ESRD; myocardial native T1 values are higher in patients with ESRD than controls, and associate with measures of myocardial strain and circulating markers of cardiac dysfunction. Although native T1 times are affected by water content of tissues, our group has shown that native T1 times are not influenced by clinical changes in fluid status in HD patients and that the inter-study reproducibility and intra- and inter-observer variability of native T1 are outstanding.

Native T1 mapping is a promising, non-invasive imaging biomarker of myocardial fibrosis in patients with advanced renal disease. It is essential that the technique is validated against histology before further use in clinical studies.

The aim of this study is to directly assess the relationship between native T1 mapping and levels of MF examined at post-mortem in haemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent haemodialysis patient (more than 3 months)
* Active on the supportive care register with anticipated death in the subsequent 12 months
* Able to give informed consent
* Consent to donation of heart for research following death
* Able to understand written and verbal explanations in English

Exclusion Criteria:

* Contraindication to MRI scan (e.g. pacemaker, incompatible metallic implants, claustrophobia)
* Patients with expected or potential infiltrative cardiomyopathy (e.g. amyloidosis)
* Unable to give informed consent
* Unable to understand written and verbal explanations in English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The plans for patient recruitment were developed in partnership with our local haemodialysis patient participation and involvement group. Patients will be identified by means of a well established supportive care register for haemodialysis patients. These patients, and often their families, have engaged in discussion about end-of-life care, including discussions about limitations on care and preferred place of death.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2019-11-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between MRI and histological measures of cardiac fibrosis | Cardiac MRI performed within 12-months of histological samples obtained post-mortem
  To assess the correlation between native T1 values measured using cardiac MRI in haemodialysis patients approaching the end of their lives, with histological samples analysed post-mortem.

SECONDARY OUTCOMES:
Accuracy of MRI versus ECHO in the measurement of cardiac fibrosis | Echocardiograms performed within 12-months of histological samples obtained post-mortem
  Relationship between integrated backscatter (measured with echocardiography) and levels of myocardial fibrosis on histology measured at post-mortem.
Relationship between cardiac fibrosis and heart rhythm | Continuous Holter recording performed within 12-months of histological samples obtained post-mortem
  Relationship between continuous Holter-monitor data and levels of myocardial fibrosis on histology measured at post-mortem.
Correlation between cardiac fibrosis and relevant circulating biomarkers | Samples collected within 12-months of histological samples obtained post-mortem
  Relationship between humoral markers of cardiac dysfunction of fibrosis and levels of myocardial fibrosis on histology measured at post-mortem
Additional cardiac MRI techniques and the measurement of cardiac fibrosis | Cardiac MRI performed within 12-months of histological samples obtained post-mortem
  The relationship between additional, non-contrast CMR techniques and histology at post-mortem

CONTACTS AND LOCATIONS:
Overall Officials: James Burton, DM, FRCP, Principal Investigator — Associate Professor in Renal Medicine
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol will be published online, open access.
Supporting Information: Study Protocol, SAP
Time Frame: The protocol will be published within 12 months of registration.
Access Criteria: Open access.